CLINICAL TRIAL: NCT01625793
Title: Inflammation, Stress and Social Behavior: Using Ecological Assessments and Model Systems to Enhance Relevance to Health Outcomes
Brief Title: Inflammation, Stress & Social Behavior: Using Ecological Assessments & Model Systems to Enhance Relevance to Health Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: New medication coming on the market, made study obsolete.
Sponsor: University of Arizona (Other)
Collaborators: Emory University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-0166-02; 5R01AT007297-03 (NIH)
Record Dates: First submitted 2012-06-11; First posted 2012-06-21 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; interferon; stress; social behavior
MeSH Terms: conditions — Hepatitis C; Social Behavior | interventions — Interferon-alpha; peginterferon alfa-2b; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HCV Interferon-alpha group (Active Comparator): Subjects receiving treatment with interferon (IFN)-alpha for chronic hepatitis C virus infection.
  Interventions: Drug: Interferon-alpha
- HCV Control Group (Placebo Comparator): Subjects delaying the start of treatment with interferon (IFN)-alpha for chronic hepatitis C virus infection by 7 weeks.
  Interventions: Drug: Interferon-alpha

INTERVENTIONS:
Drug: Interferon-alpha — Hepatitis C patients who are eligible to receive IFN-alpha treatment and enrolled in this study will be treated with pegylated IFN-alfa-2b or pegylated IFN-alfa-2a plus ribavirin at a dose of 800-1,400 mg/d as determined by the treating gastroenterologist. All medication administration is for purely clinical indications as dictated by treating physicians. Any and all diagnostic or treatment issues related to potential treatment with IFN-alpha will be conducted by treating clinicians. Subjects will be randomized to start their clinical (non-research) treatment following completion of baseline assessments or to delay the start of their clinical (non-research) treatment by 7 weeks.
  Other Names: Pegintron®, Schering Plough; PEGASYS®, Roche

SUMMARY:
The current study has been designed to identify behavioral and physiological mechanisms through which positive social connectivity (PCS) and negative social processes (NSP) interact with psychosocial stress to promote resilience in the context of illness. The investigators model inflammation (a central element of all disease states) through the use of treatment with interferon (IFN)-alpha, which provides a standardized regimen of chronic cytokine exposure known to produce profound behavioral disturbances, including depression, fatigue and sickness, in a high percentage of individuals. To objectively assess social processes, the current project will employ the Electronically Activated Recorder (EAR), which periodically and unobtrusively records snippets of ambient sounds in people's momentary environments. To objectively assess behavioral and physiological responses to psychosocial stress the current project will employ the Trier Social Stress Test (TSST), a standardized laboratory stressor known to reliably activate behavioral, neuroendocrine and inflammatory responses. These novel methodologies and model systems will be employed to test the hypotheses that (a) pre-existing affiliative and prosocial behavior will promote resilience in the context of chronic inflammation and that (b) -conversely-chronic inflammation will reduce affiliative and prosocial behavior via effects on stress reactivity, neuroendocrine function and sleep. Finally, it will explore (c) the potential mediating role of stress physiology. To test these hypotheses, 110 subjects with chronic hepatitis C virus infection will be randomized to receive treatment with pegylated IFN-alpha plus ribavirin or to postpone treatment for 6 weeks: 55 subjects at University of Arizona and 55 subjects at Emory University. Prior to randomization and 6 weeks later all subjects will be evaluated with the EAR and sleep actigraphy in their home environments and will undergo TSST and 14 hour diurnal neuroendocrine and immune measurement.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65 years including males, females and minorities
* Ability to speak and read remedial English
* Serum positive for either anti-HCV antibodies or HCV-RNA positive by PCR
* Compensated liver disease with the following minimum hematologic and biochemical criteria: hemoglobin ≥13 g/dl for males; ≥12 g/dl for females, white blood cell count > 3,000/mm3, neutrophil count >1,5000/mm3, platelets > 100,000/mm3, prothrombin time ≤ 2 seconds prolonged compared to control, or equivalent INR ratio, albumin stable and within normal limits, serum creatinine within normal limits, thyroid-stimulating hormone within normal limits, direct bilirubin ≤ 0.3 mg/dl or within 20% of upper limit of normal (ULN) for local laboratory, indirect bilirubin ≤ 0.8 mg/dl or within 20% of ULN for local laboratory, fasting blood sugar ≤ 115 mg/dl or within 20% of ULN for non-diabetic patients
* Negative pregnancy test for women of childbearing potential, and confirmation and documentation that adequate contraception or monogamous relationship with a male partner who has had a vasectomy during the treatment period and for 6 months after discontinuation of therapy
* Not breastfeeding
* Documentation and confirmation of adequate contraception in sexually active males
* Free from all psychotropic medications for 14 days prior to baseline visit (8 weeks for fluoxetine)

Exclusion Criteria:

* Evidence of untreated or poorly controlled endocrine, cardiovascular, hematological, renal, or neurological disease
* Evidence of decompensated liver disease (such as a history or presence of ascites, bleeding varices, spontaneous encephalopathy)
* History of narcolepsy, PLMS or sleep apnea (or documented during the adaptation night)
* History of CNS trauma or active seizure disorder requiring medication
* Any cause for liver disease other than chronic hepatitis C, such as co-infection with hepatitis B virus and/or human immunodeficiency virus, hemochromatosis, or Wilson's diseases
* Prior treatment with ribavirin or other antiviral or immunomodulatory drugs, including corticosteroids within 6 months of entry into protocol
* Chronic use of agents known to affect monoamine metabolism/function (and hence potentially affect the TSST), including, but not limited to, alpha- and beta-receptor agonists and antagonists, methylphenidate hydrochloride, dextroamphetamine, midodrine hydrochloride, theophylline, ephedrine, systemic antifungal azoles, sumatriptan succinate
* Psychotropic medications within 14 days prior to baseline visit (8 weeks for fluoxetine)
* Clinical gout
* Hypersensitivity to alpha interferon or ribavirin
* Hemoglobinopathies (e.g. thalassemia)
* A positive pregnancy test
* Organ transplants
* A score of <24 on the Mini Mental Status Exam (MMSE)
* Active, effective treatment of depression with an antidepressant within the past six months
* Actively meet criteria for major depression within the past six months
* Meet criteria for schizophrenia or bipolar disorder (mania) past or present
* Active abuse of alcohol or illicit/prescription drugs within the past year any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with participating in or completing the protocol

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Percent time laughing | 7 weeks
Percent time expressing empathy for others | 7 weeks
Percent of time spent in substantive conversations | 7 weeks
Percent of time spent alone | 7 weeks

SECONDARY OUTCOMES:
Cortisol concentrations in blood in response to stress test | 7 weeks
Interleukin (IL)-6 concentrations in the blood in response to stress test | 7 weeks
Diurnal plasma concentrations of interleukin-6 and tumor necrosis factor-alpha type II receptors in response to a stress test | 7 weeks
Diurnal plasma concentrations of inflamcortisol in response to a stress test | 7 weeks
Wake time after sleep onset measured by actigraphy | 7 weeks
Sleep latency by measured by actigraphy | 7 weeks
Total sleep time by actigraphy | 7 weeks
Sleep efficiency by actigraphy | 7 weeks
Structured Interview Guide for the Hamilton Depression Scale and Inventory of Depressive Symptomatology (SIGH-IDS) | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Raison, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - Emory University, Atlanta, Georgia